CLINICAL TRIAL: NCT04885114
Title: A Phase 1B, Open-label, Randomized, Controlled, Multicenter, Dose Escalation Study of the Safety, Tolerability, and Biological Effects of VY-HTT01 Administered Via Intraparenchymal Infusion of the Putamen and Thalamus in Adults With Huntington's Disease
Brief Title: Safety and Tolerability Study With VY-HTT01, in Adults With Early Manifesting Huntington's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We have discontinued our 1st generation HD program with the VYTAL Study & have initiated a 2nd generation program using a novel, proprietary AAV capsid that may enable intravenous administration & achieve widespread distribution to affected tissue.
Sponsor: Voyager Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VY-HTT01-1
Record Dates: First submitted 2021-03-02; First posted 2021-05-13 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Unilateral low dose (Experimental): 3.0 x 10^9 (vg/mL) rAAV1-miHHT
  Interventions: Genetic: Intraparenchymal rAAV1 - (mi)RNA HTT
- Cohort 2 Bilateral low dose (Experimental): 3.0 x 10^9 (vg/mL) rAAV1-miHHT
  Interventions: Genetic: Intraparenchymal rAAV1 - (mi)RNA HTT
- Cohort 3 Bilateral mid dose (Experimental): 1.7 x 10^10 (vg/mL) rAAV1-miHHT
  Interventions: Genetic: Intraparenchymal rAAV1 - (mi)RNA HTT
- Cohort 4 Bilateral high dose (Experimental): 9.9 x 10^10 (vg/mL) rAAV1-miHHT
  Interventions: Genetic: Intraparenchymal rAAV1 - (mi)RNA HTT

INTERVENTIONS:
Genetic: Intraparenchymal rAAV1 - (mi)RNA HTT — Single dose MRI guided intraparenchymal infusion of rAAV1 - (mi)RNA HTT.
  Other Names: VY-HTT01

SUMMARY:
This is the first clinical study of VY-HTT01, a gene therapy for early-stage Huntington's Disease (HD) patients. The primary goal of this trial is to evaluate the safety and tolerability of VY-HTT01. This study is a first in human study, Phase 1b, open-label, randomized, multicenter, dose escalation study with a delayed treatment control arm.

DETAILED DESCRIPTION:
This dose escalation trial will evaluate the safety and tolerability of 4 single dose levels of VY-HTT01. The maximum duration that a subject randomized to treatment may be involved in the study is up to 15 months. Delayed treatment subjects will be followed for a minimum of 6 months as a control before moving up into the treatment arm in the next cohort. The maximum duration that a delayed treatment subject may be involved in the study is up to 24 months. Subjects who participate in this study will be asked to enroll in a long-term observation study.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Have CAGn repeat >39.
* Have diagnostic confidence score of 4 based on motor, cognitive, or behavioral symptoms.
* Have a TFC score of 13 to 11.
* Have stable dosing of neurological and psychiatric medications.
* Capable of giving informed consent.
* Able to comply with all procedures and study visits.

Exclusion Criteria:

* Have any significant structural or degenerative neurologic disease other than HD.
* Have any chronic disability, significant systemic illness and/or, unstable medical condition, or clinical findings noted.
* Have primary or secondary immune-compromise due to infections or medical conditions or chronic therapies.
* Have contraindications to lumbar puncture or increased risks of bleeding upon surgery.
* Started or changed dose of a concomitant CNS medication within 30 days.
* Had prior neurosurgical procedures that could complicate the study procedures.
* Have used any investigational therapies within 30 days prior to Screening, oligonucleotide therapies within 9 months prior to Baseline, or any prior gene therapy.
* Male or female with reproductive capacity and is unwilling to use highly effective contraception for 12 months after surgery.
* Have contraindications to MRI such as claustrophobia, embedded metal in the body, or known allergy or intolerance to contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of AEs | Collected for duration of study, average of 1 year after treatment
  Safety will be assessed by measuring the number and type of AE or SAEs.

SECONDARY OUTCOMES:
Level of VY-HTT01 in blood | Collected for duration of study, average of 1 year after treatment
  Change in baseline of the levels of VY-HTT01 vector genome in blood over time.
Unified Huntington Disease Rating Scale (UHDRS) | Collected for duration of study, average of 1 year after treatment
  UHDRS will assess changes from baseline in summary scores of motor function, cognitive function, behavioral function, and functional abilities. UHDRS uses a 5-point ordinal scale ranging from 0-4 with the highest score indicating a more severe (worse) outcome.
Clinical Global Impression (CGI) Measures | Collected for duration of study, average of 1 year after treatment
  CGI-Global Improvement measure will assess changes from baseline in CGI-Severity of Illness score. Both CGI-Global Improvement and CGI- Severity measures are based on a 7-point scale, with the highest score indicating a more severe (worse) outcome.
Huntington's Disease Quality of Life (HD-QOL) Measure | Collected for duration of study, average of 1 year after treatment
  HD-QOL measure will assess changes from baseline in the HD-QOL score using a 40-question scale to identify quality of life in HD. HD-QOL is based on a 7-point scale of frequency ranging from "never" to "all of the time" with "extreme problems" indicating a more severe (worse) outcome.
EuroQol 5 Dimension 5 Level (EQ-5D-5L) Measure | Collected for duration of study, average of 1 year after treatment
  EQ-5D-5L measure will assess changes from baseline in the EQ-5D-5L score across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems", with "extreme problems" indicating a more severe (worse) outcome.

OTHER OUTCOMES:
Magnetic Resistance Imagining (MRI) | Collected for duration of study, average of 1 year after treatment
  MRI assessments will include whole brain volume, white matter volume, gray matter volume, and ventricular volume, and volumes of the putamen and thalamus covered by VY-HTT01 infusions during surgery.
Levels of HTT protein in CSF | Collected for duration of study, average of 1 year after treatment
  Change from baseline in levels of HTT protein in CSF (Cerebrospinal fluid) over time.
Levels of HTT protein in blood | Collected for duration of study, average of 1 year after treatment
  Change from baseline in levels of HTT protein in blood over time.
Huntington's Disease Cognitive Assessment Battery (HD-CAB) Measure | Collected for duration of study, average of 1 year after treatment
  HD-CAB measure will assess changes from baseline in the HD-CAB score for cognitive dysfunction in early manifest HD patients. HD-CAB consists of 6 tests; (1) Symbol Digit Modality Test (SDMT), (2) Paced Tapping, (3) One Touch Stockings of Cambridge, (4) Emotional Recognition, (5) Trial Making B and (6) Hopkins Learning Test. A multi-component score is derived by transforming the subject's score on each cognitive test to a z-score. The six z-scores are averaged to produce the HD-CAB score. A positive change from baseline indicates improvement in cognitive function; a negative change indicates worsening in cognitive function.
Level of Neurofilament Light chain (NfL) in CSF | Collected for duration of study, average of 1 year after treatment
  Change from baseline in levels of NfL in CSF over time.
Level of Neurofilament Light chain (NfL) in blood | Collected for duration of study, average of 1 year after treatment
  Change from baseline in levels of NfL in blood over time.

IPD SHARING:
Plan to Share IPD: Undecided